CLINICAL TRIAL: NCT00473525
Title: A Phase 2a, Randomized, Placebo-Controlled, Parallel Group, Multiple-Dose Study To Evaluate The Efficacy, Safety, And Tolerability Of 12-Week Oral Administration Of PF-00734200 Tablets To Subjects With Type 2 Diabetes Mellitus On Stable Treatment With Metformin
Brief Title: 12 Week Study Of PF-00734200 For The Treatment Of Type 2 Diabetes Mellitus In Subjects Treated With Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A7941005
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — gosogliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-00734200 10 mg QD (Experimental)
  Interventions: Drug: PF-00734200 10 mg QD
- PF-00734200 20 mg QD (Experimental)
  Interventions: Drug: PF-00734200 20 mg QD
- PF-00734200 5 mg QD (Experimental)
  Interventions: Drug: PF-00734200 5 mg QD
- PF-00734200 2 mg QD (Experimental)
  Interventions: Drug: PF-00734200 2 mg QD

INTERVENTIONS:
Drug: Placebo — Placebo QD
  Arms: Placebo
Drug: PF-00734200 10 mg QD — 10 mg QD
  Arms: PF-00734200 10 mg QD
Drug: PF-00734200 20 mg QD — 20 mg QD
  Arms: PF-00734200 20 mg QD
Drug: PF-00734200 5 mg QD — 5 mg QD
  Arms: PF-00734200 5 mg QD
Drug: PF-00734200 2 mg QD — 2 mg QD
  Arms: PF-00734200 2 mg QD

SUMMARY:
The purpose of this Phase 2a study is to evaluate the efficacy, safety and tolerability, of multiple parallel doses of PF-00734200 following oral administration to adult human subjects with T2DM who currently are on a stable dose of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Hb1AC >7%-11% inclusive
* Male and females 18-70; females must be post-menopausal
* On a stable dose of metformin hydrochloride

Exclusion Criteria:

* Medical history of stroke, unstable angina, heart attack within one year of enrollment, and alcohol dependency or recent drug abuse.
* Women of childbearing potential, pregnant or nursing
* Evidence of diabetic complications with significant end-organ damage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
HbA1C levels (%) | 12 weeks
Evaluation of Dose Response in HbA1c (%) | 12 weeks

SECONDARY OUTCOMES:
Insulin and Glucose AUC following a mixed meal tolerance test | 12 weeks
Proportion of subjects achieving ADA glycemic goal of Hb A1c <7% | 12 weeks
Incidence of Adverse Events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (65):
- United States (52):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Carmichael, California
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, Fair Oaks, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Roseville, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, DeFuniak Springs, Florida
  - Pfizer Investigational Site, Destin, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Skokie, Illinois
  - Pfizer Investigational Site, Wheeling, Illinois
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Brockton, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Canton, Michigan
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Biloxi, Mississippi
  - Pfizer Investigational Site, Picayune, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Trenton, New Jersey
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Marion, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Carnegie, Pennsylvania
  - Pfizer Investigational Site, East Providence, Rhode Island
  - Pfizer Investigational Site, Bartlett, Tennessee
  - Pfizer Investigational Site, Collierville, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Colombia (2):
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Floridablanca, Santander Department
- Germany (4):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Giengen an der Brenz
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, München
- Pfizer Investigational Site, Roma, Italy
- Spain (3):
  - Pfizer Investigational Site, Santiago de Compostela, La Coruña
  - Pfizer Investigational Site, Alcalá de Henares, Madrid
  - Pfizer Investigational Site, Valencia, Valencia
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Stockholm

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7941005&StudyName=12%20Week%20Study%20Of%20PF-00734200%20For%20The%20Treatment%20Of%20Type%202%20Diabetes%20Mellitus%20In%20Subjects%20Treated%20With%20Metformin